CLINICAL TRIAL: NCT07101029
Title: Effect of Bio-C Temp Versus Calcium Hydroxide as an Intracanal Dressing on Postoperative Pain Intensity and Periapical MMP-9 Level in Patients With Necrotic Pulp: A Randomized Clinical Trial
Brief Title: Effect of Bio-C Temp Versus Calcium Ydroxide as Intracanal Dressings on Postoperative Pain Intensity and Periapical MMP-9 Level in Patients With Necrotic Pulp
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Alaa El-Dien Mohamed, Assisstant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MennaalaaCU25
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Intracanal Dressing; Apical Periodontitis; Calcium Hydroxide; Biomarkers; Inflammatory Mediators
Keywords: Bio-C Temp; Calcium Hydroxide; Intracanal medicament; Matrix Metalloproteinase 9; Biomarkers; Post operative pain
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-C Temp (Experimental): This group will Receive Bio-C Temp Bioceramic paste as intracanal dressing
  Interventions: Drug: Bio-C Temp Intracanal Medication
- Calcium Hydroxide (Active Comparator): This group will Receive Calcium Hydroxide paste as intracanal dressing
  Interventions: Drug: Calcium Hydroxide Intracanal medication

INTERVENTIONS:
Drug: Bio-C Temp Intracanal Medication — Bio-C Temp Bioceramic intracanal dressing in the form of injectable premixed paste
  Other Names: Bioceramic intracanal dressing
  Arms: Bio-C Temp
Drug: Calcium Hydroxide Intracanal medication — Calcium Hydroxide intracanal dressing in the form of injectable premixed paste
  Arms: Calcium Hydroxide

SUMMARY:
To compare the effect of Bio-C Temp Bioceramic intracanal dressing versus calcium hydroxide as intracanal medicaments on:

* Intensity of postoperative pain
* levels of MMP -9 in Periapical Fluids.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-50 years old.
2. Males and females.
3. Healthy patients categorized as I or II according to The American Society of Anesthesiologists.

   (ASA I or II), with no underlying allergies.
4. Single-rooted mandibular premolar teeth, having single root canal:

   * Diagnosed clinically with pulp necrosis.
   * Absence of spontaneous pulpal pain.
   * Slight widening in the periodontal membrane space or with periapical radiolucency not exceeding 2*2 mm radiographically.
5. Patients accepting to participate in the trial.
6. Patients who can understand pain scale and can sign the informed consent

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders (ASA III or IV).
2. Pregnant females.
3. If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively as it might alter their pain perception.
4. Teeth with multiple canals. 9
5. Teeth that show association with acute periapical abscess, swelling or fistulous tract.
6. Teeth with vital pulp.
7. Non-restorable teeth or teeth that could not be adequately isolated with a rubber dam.
8. Immature teeth.
9. Teeth with greater than grade I mobility or pocket depth greater than 4 mm.
10. Teeth showing radiographic evidence of external or internal root resorption, vertical root fracture, perforation or calcification.
11. Patients with two or more adjacent teeth requiring endodontic treatment.
12. Patients reporting bruxism, clenching or TMJ problems.
13. Inability to perceive the given instructions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intensity of post-operative pain | 6 hours post-instrumentation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 12 hours post-instrumentation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 24 hours post-instrumentation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 48 hours post-instrumentation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 6 hours post-obturation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 12 hours post-obturation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 24 hours post-obturation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)
Intensity of post-operative pain | 48 hours post-obturation
  Intensity of post-operative pain as measured by Numerical Rating Scale (NRS)

SECONDARY OUTCOMES:
Periapical MMP-9 level | at the first visit post- instrumentation
  Level Of MMP-9 Enzyme in the periapical tissue fluid, quantified by ELISA
Periapical MMP-9 Level | After 1 week at the second visit (pre-obturation)
  Level of MMP-9 enzyme in the periapical tissue fluid, Quantified by ELISA